CLINICAL TRIAL: NCT03218748
Title: Adaptation and Evaluation of the Honest, Open, Proud Program for Soldiers with Mental Illness
Brief Title: Honest, Open, Proud for Soldiers with Mental Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulm (Other)
Collaborators: Center for Military Mental Health, Berlin, Germany (Unknown); Illinois Institute of Technology, Chicago, USA (Unknown)
Responsible Party: Principal Investigator, Nicolas Rüsch, Professor, University of Ulm
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HOP Soldiers
Record Dates: First submitted 2017-07-12; First posted 2017-07-17 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Mental Illness
Keywords: Mental illness; Disclosure; stigma; soldiers; secrecy
MeSH Terms: conditions — Mental Disorders; Social Stigma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Honest, Open, Proud (Experimental): The group program is about disclosure versus secrecy of one's mental illness. The groups are facilitated by two peers (soldiers with lived experience of mental illness). Each group runs for three weeks, one meeting per week, and two hours per meeting. There is one 2-hour booster session in week 6.
  Fidelity to manual: rated by a research assistant who is present during the group session
  Interventions: Behavioral: Honest, Open, Proud (HOP)
- Control group (No Intervention): Treatment as usual (TAU)

INTERVENTIONS:
Behavioral: Honest, Open, Proud (HOP) — Three lessons, one for each two-hour session plus one booster session
  1. Considering the pros and cons of disclosure:
     Discussion of one's idea of identity and mental illness, weighing the costs and benefits of (non-) disclosure
  2. Different ways to disclose:
     Discussion of different levels of (non-) disclosure, considering costs and benefits of each level, selecting persons to disclose to and how to test them out, anticipating responses of others to one's disclosure
  3. Telling one's story:
     Practice how to tell one's story, identifying peers who might be helpful with the coming out process
  4. Booster session Reviewing previous intentions to disclose one's mental illness, discussion whether one disclosed and evaluating this experience
  Other Names: Coming Out Proud (COP)
  Arms: Honest, Open, Proud

SUMMARY:
The purpose of the study is to evaluate the feasibility and efficacy of the group-based intervention "Honest, Open, Proud" among soldiers with mental illness.

DETAILED DESCRIPTION:
Soldiers with mental illness typically face a two-fold problem. On the one hand, they have to cope with the symptoms of their mental illness; on the other hand, they often have to deal with stigma and discrimination. Both due to fear of public stigma and due to self-stigma or shame, soldiers with mental illness may decide to keep their condition a secret or even to withdraw from other people altogether in order to minimize the risk of being labeled. Secrecy can help on the short term to protect individuals from public stigma, but usually it has negative long-term consequences such as social isolation, distress and avoidance of help-seeking. Disclosure, on the other hand, carries the risk to be discriminated by others, but can reduce the burden of secrecy, lead to support by others and reduce public stigma.

In this study investigators aim to test the efficacy (see our outcomes above) of Honest, Open, Proud run by soldiers with lived experience of mental illness.

ELIGIBILITY:
Inclusion Criteria:

* At least one self-reported current axis I or axis II disorder according to DSM-5, which is not restricted to only substance-related disorder(s)
* Age 18 or above
* Ability to provide written informed consent
* Fluent in German (needed for self-report measures)
* At least a moderate level of self-reported disclosure-related distress/difficulty (score 4 or higher on the screening item 'In general, how distressed or worried are you in terms of secrecy or disclosure of your mental illness to others?', rated from 1, not at all, to 7, very much)
* Current inpatient, day-clinic or outpatient treatment at the Center for Military Mental Health, Berlin, Germany
* from April 2018 onwards we decided to also include non-military first responders (fire fighters or police officers) who are treated in the Center for Military Mental Health, Berlin, Germany

Exclusion Criteria:

* Self-reported diagnosis of only a substance- or alcohol-related disorder, without non-substance related current psychiatric comorbidity. We will exclude people who only have a substance-/alcohol-related disorder because the disclosure of these disorders is not the topic of the HOP intervention
* Intellectual disability
* Organic disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Stigma Stress Scale, 8 items | 3 weeks (T1)
  (Rüsch et al. 2009a; Rüsch et al. 2009b)
WHOQoL BREF; Domain psychological quality of life, 6 items | 6 weeks (T2)
  (WHOQoL Group 1998)

SECONDARY OUTCOMES:
Empowerment Scale, Subscale 'Self-esteem', 9 items | baseline, 3, 6 and 12 weeks (T3)
  (Rogers et al. 1997)
Psychological Well-Being Scale, 18 items | baseline, 3, 6 and 12 weeks
  (Ryff 1989)
Internalized Stigma of Mental Illness Inventory, Brief Version, 10 items | baseline, 3, 6 and 12 weeks
  (Boyd et al. 2014)
Self-Stigma of Mental Illness Scale, Short Version, subscale Self-Concurrence, 5 items | baseline, 3, 6 and 12 weeks
  (Corrigan et al. 2012)
Secrecy and Social Withdrawal subscales of the Stigma Coping Orientation Scales, 12 items | baseline, 3, 6 and 12 weeks
  (Link et al. 1991)
Disclosure related distress ("In general, how distressed or worried are you in terms of secrecy or disclosure of your mental illness to others?', from 1, not at all, to 7, very much) | baseline, 3, 6 and 12 weeks
  (Rüsch et al. 2014a)
WHOQoL-BREF, 26 items | 3, 6 and 12 weeks
  (WHOQOL Group 1998)
Patient Health Questionnaire (PHQ-9), 9 items | baseline, 3, 6 and 12 weeks
  (Kroenke et al. 2001)
Shame about having a mental illness, 1 item | baseline, 3, 6 and 12 weeks
  (Rüsch et al. 2014b)
Attitudes to help-seeking, 2 items | baseline, 3, 6 and 12 weeks
  (Rüsch et al. 2013)
Attitudes to disclosure, 2 items | baseline, 3, 6 and 12 weeks
  (Rüsch et al. 2011)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Rüsch, Dr., Principal Investigator — Department of Psychiatry II, Section Public Mental Health, Ulm University, Bezirkskrankenhaus Günzburg; Gerd-Dieter Willmund, Dr., Principal Investigator — Center for Military Mental Health, Berlin, Germany; Peter Zimmermann, Dr., Principal Investigator — Center for Military Mental Health, Berlin, Germany
Locations (3):
- Illinois Institute of Technology, Chicago, Illinois, United States
- Germany (2):
  - Center for Military Mental Health, Berlin
  - Department of Psychiatry II, Section Pubic Mental Health, Ulm University, Bezirkskrankenhaus Günzburg, Ulm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rogers ES, Chamberlin J, Ellison ML, Crean T. A consumer-constructed scale to measure empowerment among users of mental health services. Psychiatr Serv. 1997 Aug;48(8):1042-7. doi: 10.1176/ps.48.8.1042. PMID 9255837
- [Background] Boyd JE, Otilingam PG, Deforge BR. Brief version of the Internalized Stigma of Mental Illness (ISMI) scale: psychometric properties and relationship to depression, self esteem, recovery orientation, empowerment, and perceived devaluation and discrimination. Psychiatr Rehabil J. 2014 Mar;37(1):17-23. doi: 10.1037/prj0000035. PMID 24660946
- [Background] Corrigan PW, Michaels PJ, Vega E, Gause M, Watson AC, Rusch N. Self-stigma of mental illness scale--short form: reliability and validity. Psychiatry Res. 2012 Aug 30;199(1):65-9. doi: 10.1016/j.psychres.2012.04.009. Epub 2012 May 10. PMID 22578819
- [Background] Rusch N, Abbruzzese E, Hagedorn E, Hartenhauer D, Kaufmann I, Curschellas J, Ventling S, Zuaboni G, Bridler R, Olschewski M, Kawohl W, Rossler W, Kleim B, Corrigan PW. Efficacy of Coming Out Proud to reduce stigma's impact among people with mental illness: pilot randomised controlled trial. Br J Psychiatry. 2014;204(5):391-7. doi: 10.1192/bjp.bp.113.135772. Epub 2014 Jan 16. PMID 24434073
- [Background] Link BG, Mirotznik J, Cullen FT. The effectiveness of stigma coping orientations: can negative consequences of mental illness labeling be avoided? J Health Soc Behav. 1991 Sep;32(3):302-20. PMID 1940212
- [Background] Rusch N, Corrigan PW, Heekeren K, Theodoridou A, Dvorsky D, Metzler S, Muller M, Walitza S, Rossler W. Well-being among persons at risk of psychosis: the role of self-labeling, shame, and stigma stress. Psychiatr Serv. 2014 Apr 1;65(4):483-9. doi: 10.1176/appi.ps.201300169. PMID 24382666
- [Background] Rusch N, Heekeren K, Theodoridou A, Dvorsky D, Muller M, Paust T, Corrigan PW, Walitza S, Rossler W. Attitudes towards help-seeking and stigma among young people at risk for psychosis. Psychiatry Res. 2013 Dec 30;210(3):1313-5. doi: 10.1016/j.psychres.2013.08.028. Epub 2013 Sep 4. PMID 24012162
- [Background] Rusch N, Evans-Lacko SE, Henderson C, Flach C, Thornicroft G. Knowledge and attitudes as predictors of intentions to seek help for and disclose a mental illness. Psychiatr Serv. 2011 Jun;62(6):675-8. doi: 10.1176/ps.62.6.pss6206_0675. PMID 21632739
- [Background] Development of the World Health Organization WHOQOL-BREF quality of life assessment. The WHOQOL Group. Psychol Med. 1998 May;28(3):551-8. doi: 10.1017/s0033291798006667. PMID 9626712
- [Background] Rusch N, Corrigan PW, Powell K, Rajah A, Olschewski M, Wilkniss S, Batia K. A stress-coping model of mental illness stigma: II. Emotional stress responses, coping behavior and outcome. Schizophr Res. 2009 May;110(1-3):65-71. doi: 10.1016/j.schres.2009.01.005. Epub 2009 Feb 23. PMID 19237266
- [Background] Rusch N, Corrigan PW, Wassel A, Michaels P, Olschewski M, Wilkniss S, Batia K. A stress-coping model of mental illness stigma: I. Predictors of cognitive stress appraisal. Schizophr Res. 2009 May;110(1-3):59-64. doi: 10.1016/j.schres.2009.01.006. Epub 2009 Mar 6. PMID 19269140
- [Background] Ryff, C. D. (1989): Happiness is everything, or is it? Explorations on the meaning of psychological well-being. Journal of Personality and Social Psychology (57): 1069-1081.
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Derived] Rusch N, Helms C, Horger J, Hohle B, Bernert H, Muschner P, Rose C, Corrigan PW, Mulfinger N, Zimmermann P, Willmund GD. The peer-led Honest, Open, Proud program to decrease the impact of mental illness stigma among German military personnel: randomized controlled trial. Soc Psychiatry Psychiatr Epidemiol. 2025 Jul 22. doi: 10.1007/s00127-025-02960-x. Online ahead of print. PMID 40696200